CLINICAL TRIAL: NCT02038491
Title: RICALOR - Registro Italiano Complicanze Anestesia LOco Regionale - Italian Registry for Complications During Regional Anesthesia
Brief Title: RICALOR Italian Registry for Complications During Regional Anesthesia
Acronym: RICALOR
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 20090016600; PT SM 05 Ricalor (Other: Policlinico S Matteo Pavia Italy)
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Spinal Hematoma; Spinal Abscess; Neurologic Manifestations; Cardiovascular Diseases; Respiratory Failure
Keywords: Epidural anesthesia; Spinal anesthesia; nerve blocks; complications
MeSH Terms: conditions — Neurologic Manifestations; Cardiovascular Diseases; Respiratory Insufficiency | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- regional anesthesia: patients undergoing regional anesthesia procedures
  Interventions: Procedure: regional anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — Spinal, epidural, combined spinal epidural, nerve blocks

SUMMARY:
Regional anesthesia is the cornerstone of modern postoperative analgesia, but concerns remain about possible adverse effects and complication.

RICALOR Group Investigators developed a national registry to register the incidence of regional anesthesia-associated complications and to identify possible risk factors.

DETAILED DESCRIPTION:
The project has been advertised through direct contact with relevant organizations in anaesthesia and pain management. Any other center willing to participate is provided with all the documents to receive its local Institutional Review Board (IRB) approval, and a 'local responsible' (LR) is nominated to co-ordinate the project and to be responsible of data collection locally.

Centers receiving IRB approval collect data about different types of procedure (adult major and minor surgery, pediatric surgery, obstetric anesthesia, pain management). Data are collected on a specifically designed form, and every center quarterly sent the promoter centre a report including general data and a specific report for every occurred complication.

Eligibility criteria

Investigators collect the total number of intervention and the number of regional anesthesia(RA) techniques performed . Patients recorded as "case" and "controls" had to sign a specifical informed consent. For pediatric patients and patients not able to sign for any reason, a specific form is included in the document, to be signed by parents or any legally-established tutor, as required for every clinical procedure or scientific trial in our country.

General data

Total number of interventions, the number of central neuraxial block (CNBs), peripheral nerve blocks (PNBs) and continuous PNBs (CPNBs) performed. CNBs are classified as epidurals, combined spinal-epidurals (CSEs), subarachnoid. PNBs and cPNBs are divided into ultrasound-guided, nerve stimulation-guided and blind techniques.

Specific data - report for complications

For each complication a specific report is sent for data analysis, including data concerning cases (patient with complication) and controls (the two following patients undergoing the same type of loco-regional technique).

Reports are slightly different for CNBs and (c)PNBs. For every patient, the investigators register demographic data (age, ASA-American Society of Anesthesiologists- status, height and weight), data regarding surgical technique (type of surgery, open/video-laparoscopic/robotic approach, election/emergency surgery) and data regarding anti-thromboembolic therapy (drugs, timing of suspension before/after blockade).

A second part of the report is strictly dedicated to the technique and to the type of complication occurred (and, hence, different in central and peripheral blocks).

Statistical analysis

Study population is estimated basing on previous studies of major complications after CNBs, which indicate an incidence of major adverse effects of 4.2 on 100.000 patients. Estimating an incidence of 1:25.000, a number of 25.000 procedures was calculated to be needed for the study, with a confidence interval of 95%. The primary endpoint was to assess cumulative incidence of adverse effects, while a following case-control analysis will be performed to identify possible risk factors.

ELIGIBILITY:
Inclusion Criteria:

* M/F
* undergoing surgery or procedures needing regional anesthesia
* signed informed consent for data treatment

Exclusion Criteria:

* no informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing surgery with regional anesthesia during study period will be considered for complications' incidence calculation .
Sampling Method: Probability Sample
Enrollment: 63692 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
number of subjects presenting complications associated with regional anesthesia techniques | 6 months
  Number of subjects presenting complications associated with regional anesthesia is recorded, and when a neurologic deficit could occur, we monitor the patient for at least 6 months

SECONDARY OUTCOMES:
statistically significant difference in cases (complication) and controls regarding factors potentially affecting complications' occurrence | up to dismission
  Case control analysis to identify risk factors connected with major complications. Analyzed variables will be: demographic variables, emergency/election surgery, equipment (needles, type of guidance), tourniquet, patients position, drugs dosing regimen, anti-thrombotic therapy, type of surgery, operator experience, type of block.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S Matteo, Pavia, Italy

REFERENCES:
- [Background] Bugada Dario; Allegri Massimo; RICALOR Group investigators; Zadra Nicola; Braschi Antonio ; Borghi Battista; Grossi Paolo.
- See also: Related Info — http://www.esraitalia.it